CLINICAL TRIAL: NCT01309932
Title: A Phase 2B, Randomized Study to Evaluate the Safety and Efficacy of Pegylated Interferon Lambda (BMS-914143) Administered With Ribavirin Plus a Single Direct Antiviral Agent (BMS-790052 or BMS-650032) Versus Pegasys Administered With Ribavirin (Part A) and of Pegylated Interferon Lambda (BMS-914143) Administered With or Without Ribavirin Plus 2 Direct Antiviral Agents (BMS-790052 and BMS-650032) (Part B) in Chronic Hepatitis C Genotype-1 Treatment naïve Subjects
Brief Title: Safety Study of Pegylated Interferon Lambda Plus Single or 2 Direct Antiviral Agents With Ribavirin
Acronym: D-LITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI452-008; 2010-022568-11 (EudraCT Number)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a; daclatasvir; Ribavirin; asunaprevir; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- A1: pegIFNλ+BMS-790052+Placebo for BMS-650032+Ribavirin (Experimental): Part A
  Interventions: Biological: Pegylated Interferon Lambda (pegIFNλ); Drug: BMS-790052 (NS5A Inhibitor); Drug: Ribavirin (RBV); Drug: Placebo (PBO) for BMS-650032 (Placebo for NS3 Protease Inhibitor)
- A2: pegIFNλ+BMS-650032+Placebo for BMS-790052+Ribavirin (Experimental): Part A
  Interventions: Biological: Pegylated Interferon Lambda (pegIFNλ); Drug: Ribavirin (RBV); Drug: BMS-650032 (NS3 Protease Inhibitor); Drug: Placebo (PBO) for BMS-790052 (Placebo for NS5A Inhibitor)
- A3: pegIFNα-2a+PBO for BMS-790052+PBO for BMS-650032+RBV (Active Comparator): Part A
  Interventions: Drug: Ribavirin (RBV); Biological: Pegylated Interferon Alfa-2a (pegIFNα-2a); Drug: Placebo (PBO) for BMS-650032 (Placebo for NS3 Protease Inhibitor); Drug: Placebo (PBO) for BMS-790052 (Placebo for NS5A Inhibitor)
- A4: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (24 weeks) (Experimental): Part B
  Interventions: Drug: BMS-790052 (NS5A Inhibitor); Drug: BMS-650032 (NS3 Protease Inhibitor); Biological: Pegylated Interferon Lambda (pegIFNλ); Drug: Ribavirin (RBV)
- A5: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (16 weeks) (Experimental): Part B
  Interventions: Biological: Pegylated Interferon Lambda (pegIFNλ); Drug: Ribavirin (RBV); Drug: BMS-790052 (NS5A Inhibitor); Drug: BMS-650032 (NS3 Protease Inhibitor)
- A6: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (24 weeks) (Experimental): Part B
  Interventions: Drug: BMS-790052 (NS5A Inhibitor); Drug: BMS-650032 (NS3 Protease Inhibitor); Biological: Pegylated Interferon Lambda (pegIFNλ); Drug: Placebo for Ribavirin (RBV)
- A7: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (16 weeks) (Experimental): Part B
  Interventions: Biological: Pegylated Interferon Lambda (pegIFNλ); Drug: BMS-790052 (NS5A Inhibitor); Drug: BMS-650032 (NS3 Protease Inhibitor); Drug: Placebo for Ribavirin (RBV)

INTERVENTIONS:
Biological: Pegylated Interferon Lambda (pegIFNλ) — Solution, Subcutaneous, 180 μg/mL, Once weekly, 24 or 48 weeks depending on response
  Other Names: BMS-914143
  Arms: A1: pegIFNλ+BMS-790052+Placebo for BMS-650032+Ribavirin; A2: pegIFNλ+BMS-650032+Placebo for BMS-790052+Ribavirin
Drug: BMS-790052 (NS5A Inhibitor) — Tablets, Oral, 60 mg, Once daily, 24 weeks
  Other Names: BMS-790052
  Arms: A1: pegIFNλ+BMS-790052+Placebo for BMS-650032+Ribavirin; A4: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (24 weeks); A6: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (24 weeks)
Drug: Ribavirin (RBV) — Tablets, Oral, 1000 or 1200 mg based on weight, Twice daily, 48 weeks
  Other Names: Ribasphere
  Arms: A1: pegIFNλ+BMS-790052+Placebo for BMS-650032+Ribavirin; A2: pegIFNλ+BMS-650032+Placebo for BMS-790052+Ribavirin; A3: pegIFNα-2a+PBO for BMS-790052+PBO for BMS-650032+RBV
Drug: BMS-650032 (NS3 Protease Inhibitor) — Tablets, Oral, 200 mg, Twice daily, 24 weeks
  Other Names: BMS-650032
  Arms: A2: pegIFNλ+BMS-650032+Placebo for BMS-790052+Ribavirin; A4: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (24 weeks); A6: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (24 weeks)
Biological: Pegylated Interferon Alfa-2a (pegIFNα-2a) — Solution, Subcutaneous, 180 μg/mL, Once weekly, 48 weeks
  Other Names: Pegasys®
  Arms: A3: pegIFNα-2a+PBO for BMS-790052+PBO for BMS-650032+RBV
Biological: Pegylated Interferon Lambda (pegIFNλ) — Solution, Subcutaneous, 180 μg/mL, Once weekly, 24 weeks
  Other Names: BMS-914143
  Arms: A4: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (24 weeks); A6: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (24 weeks)
Drug: Ribavirin (RBV) — Tablets, Oral, 1000 or 1200 mg based on weight, Twice daily, 24 weeks
  Other Names: Ribasphere
  Arms: A4: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (24 weeks)
Biological: Pegylated Interferon Lambda (pegIFNλ) — Solution, Subcutaneous, 180 μg/mL, Once weekly, 16 weeks
  Other Names: BMS-914143
  Arms: A5: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (16 weeks); A7: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (16 weeks)
Drug: Ribavirin (RBV) — Tablets, Oral, 1000 or 1200 mg based on weight, Twice daily, 16 weeks
  Other Names: Ribasphere
  Arms: A5: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (16 weeks)
Drug: BMS-790052 (NS5A Inhibitor) — Tablets, Oral, 60 mg, Once daily, 16 weeks
  Other Names: BMS-790052
  Arms: A5: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (16 weeks); A7: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (16 weeks)
Drug: BMS-650032 (NS3 Protease Inhibitor) — Tablets, Oral, 200 mg, Twice daily, 16 weeks
  Other Names: BMS-650032
  Arms: A5: pegIFNλ+BMS-790052+BMS-650032+Ribavirin (16 weeks); A7: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (16 weeks)
Drug: Placebo (PBO) for BMS-650032 (Placebo for NS3 Protease Inhibitor) — Tablets, Oral, 0 mg, Twice daily, 24 weeks
  Other Names: Placebo for BMS-650032
  Arms: A1: pegIFNλ+BMS-790052+Placebo for BMS-650032+Ribavirin; A3: pegIFNα-2a+PBO for BMS-790052+PBO for BMS-650032+RBV
Drug: Placebo (PBO) for BMS-790052 (Placebo for NS5A Inhibitor) — Tablets, Oral, 0 mg, Once daily, 24 weeks
  Other Names: Placebo for BMS-790052
  Arms: A2: pegIFNλ+BMS-650032+Placebo for BMS-790052+Ribavirin; A3: pegIFNα-2a+PBO for BMS-790052+PBO for BMS-650032+RBV
Drug: Placebo for Ribavirin (RBV) — Tablets, Oral, 0 mg, Twice daily, 24 weeks
  Other Names: Placebo for Ribasphere
  Arms: A6: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (24 weeks)
Drug: Placebo for Ribavirin (RBV) — Tablets, Oral, 0 mg, Twice daily, 16 weeks
  Other Names: Placebo for Ribasphere
  Arms: A7: pegIFNλ+BMS-790052+BMS-650032+Placebo for RBV (16 weeks)

SUMMARY:
The purpose of this study is to determine if combination therapy with Pegylated Interferon Lambda (BMS-914143) plus Ribavirin (RBV) with a single direct antiviral agent (BMS-790052 or BMS-650032) for 24 weeks is effective and safe for treatment of Chronic Hepatitis C (CHC) compared to current standard therapy with Pegylated Interferon Alpha-2a plus RBV for 48 weeks.

DETAILED DESCRIPTION:
Study Classification: Pharmacokinetics/ Pharmacodynamics

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Chronic Hepatitis C, Genotype 1
* HCV RNA >100,000 IU/mL at screening;
* Seronegative for Human immunodeficiency virus (HIV) and Hepatitis B surface antigen (HBsAg);
* Liver biopsy within prior 2 years; subjects with compensated cirrhosis can enroll and will be capped at approximately 10%

Exclusion Criteria:

* Any evidence of liver disease other than HCV;
* Co-infection with HIV;
* Diagnosed or suspected hepatocellular carcinoma;
* Medical history or laboratory value abnormalities that would prohibit the use of Pegylated Interferon Alpha-2a or Ribavirin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (as measured by the frequency of serious adverse events (SAEs), dose reductions and discontinuations due to adverse events (AEs) | Up to end of treatment ( maximum of 48 weeks) plus 30 days
Antiviral activity as determined by the proportion of Hepatitis C virus (HCV) genotype 1 subjects with 24-week sustained virologic response (SVR24) | At end of treatment (maximum of 48 weeks)
Antiviral activity as determined by the proportion of Hepatitis C virus (HCV) genotype 1 subjects with 24-week sustained virologic response (SVR24) | Post-treatment Week 24

SECONDARY OUTCOMES:
Proportion of HCV genotype 1 subjects with Protocol definition of virologic response (PDR) for Part A and Part B | Weeks 4, Weeks 12 and post-treatment Weeks 24
  * Part A PDR is defined as HCV RNA at Week 4 < LLOQ and Week 12 undetectable
  * Part B PDR is defined as HCV RNA at Week 2 ≥ 2 log10 decrease (or < Lower limit of quantitation (LLOQ) if baseline HCV RNA < 2400 IU/mL), Week 4 < LLOQ and Week 12 undetectable
Proportion of subjects with either a 2-log or greater decrease in Hepatitis C virus (HCV) Ribonucleic acid (RNA) levels from baseline or undetectable levels of HCV RNA | Weeks 2, Weeks 4 and Weeks 12
Proportion of subjects with viral breakthrough, defined as confirmed > 1 log10 increase in HCV RNA over nadir or confirmed HCV RNA ≥ Lower limit of quantitation (LLOQ) after confirmed undetectable HCV RNA while on treatment | Post-treatment Week 48
Proportion of subjects with undetectable HCV RNA at the end of treatment that develop detectable levels of HCV RNA in the post-treatment follow-up period | Post-treatment Week 48
Serum HCV Ribonucleic acid (RNA) levels over time | Days 1, 3, Weeks 1, 2, 4, 6, 8, 12, 16, 20, and end of treatment (Week 16, 24 or 48 depending on treatment assignment)
Proportion of subjects with undetectable HCV RNA over time | Days 1, 3, Weeks 1, 2, 4, 6, 8, 12, 16, 20, and end of treatment (Week 16, 24 or 48 depending on treatment assignment)
Time to viral clearance, defined as an absence of detectable HCV RNA | Day 1, 3, Week 1, 2, 4, 6, 8, 12, 24, 36, end of treatment (Week 48), Post-Treatment at Week 4, 12, 24, 36, 48, and 56
Serum levels of pegIFNλ and pegIFNα-2a and plasma levels of BMS-790052 and BMS-650032: In PK sub-study group Maximum observed serum/plasma concentration (Cmax) | Cmax will be determined at Dose 5 (Study Visit Week 4: 0 - 12 h for BMS-650032, 0 - 24 h for BMS-790052, and 0 - 168 h for pegIFNλ and pegIFNα-2a)
Serum levels of pegIFNλ and pegIFNα-2a and plasma levels of BMS-790052 and BMS-650032: In PK sub-study group Time to maximum concentration (Tmax) | Tmax will be determined at Dose 5 (Study Visit Week 4: 0 - 12 h for BMS-650032, 0 - 24 h for BMS-790052, and 0 - 168 h for pegIFNλ and pegIFNα-2a)
Serum levels of pegIFNλ and pegIFNα-2a and plasma levels of BMS-790052 and BMS-650032: In PK sub-study group Minimal observed serum/plasma concentration (Cmin) | Cmin will be determined at Dose 5 (Study Visit Week 4: 0 - 12 h for BMS-650032, 0 - 24 h for BMS-790052, and 0 - 168 h for pegIFNλ and pegIFNα-2a)
Serum levels of pegIFNλ and pegIFNα-2a and plasma levels of BMS-790052 and BMS-650032: In PK sub-study group Area under the serum/plasma concentration-time curve during one dose interval AUC(TAU) | AUC(TAU) will be determined at Dose 5 (Study Visit Week 4: 0 - 12 h for BMS-650032, 0 - 24 h for BMS-790052, and 0 - 168 h for pegIFNλ and pegIFNα-2a)
Serum levels of pegIFNλ and pegIFNα-2a and plasma levels of BMS-790052 and BMS-650032: In all subjects, trough concentrations will be assessed (Ctrough) | Troughs at baseline (week 0), weeks 2, 4, 8, 12, 16, and 24
Proportion of subjects with 12-week sustained virologic response (SVR12), defined as undetectable HCV RNA | At end of treatment (maximum of 48 weeks) and follow-up Week 12
Proportion of subjects with 4-week sustained virologic response (SVR4), defined as undetectable HCV RNA | At end of treatment (maximum of 48 weeks) and follow-up Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (39):
- United States (13):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Desert Medical Group Inc., Palm Springs, California
  - University Of Colorado Denver And Hospital, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Johns Hopkins University, Lutherville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Bristol-Myers Squibb/David E. Bernstein, Md, Manhasset, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - St. Luke'S Episcopal Hospital - Baylor College Of Medicine, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (4):
  - Local Institution, Adelaide, South Australia
  - Local Institution, Clayton Vic, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Perth, Western Australia
- France (5):
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Paris
- Germany (3):
  - Local Institution, Essen
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
- Italy (2):
  - Local Institution, Pisa
  - Local Institution, Roma
- Japan (7):
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kawasaki-shi, Kanagawa
  - Local Institution, Osaka, Osaka
  - Local Institution, Iruma-gun, Saitama
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
- New Zealand (2):
  - Local Institution, Grafton, Auckland
  - Local Institution, Christchurch
- Fundacion De Investigacion De Diego, San Juan, Puerto Rico
- Spain (2):
  - Local Institution, Barcelona, Barcelona
  - Local Institution, Valencia

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx